CLINICAL TRIAL: NCT02046954
Title: Retrospective Matched Pair Analyses for Evaluating the Influence of Hemodynamically Focussed Transesophageal Echocardiography (hTEE) on Postoperative Outcome in Cardiosurgery Patients
Brief Title: EVENT - Evaluation of the Influence of hTEE
Acronym: EVENT
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Sander, Univ.-Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: EA1/249/13
Record Dates: First submitted 2014-01-19; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Postoperative Heart Insufficiency
Keywords: transesophageal echocardiography; tee; toe; cardiac surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: Patients monitored with hemodynamically focussed transesophageal echocardiography (placement within 12 hours of ICU admission)
- Control Group: Patients receiving conventional monitoring (e.g. transpulmonary thermodilution)

SUMMARY:
Compromised tissue oxygenation during surgery may negatively influence patient outcome. Primary cause of insufficient tissue oxygenation is reduced cardiac output due to hypovolemia and/or reduced cardiac contractility. In cardiac surgery patients especially, postoperative pericardia effusion and/or tamponade may further compromise cardiac function. Today, hemodynamically instable patients are often monitored by means of pulmonal artery catheters or transpulmonary thermodilution. However, these methods only allow quantification of functional limitations. Underlying causes may be investigated by relatively recent technology through hemodynamically focussed transesophageal echocardiography (ClariTEE(R) ImaCor) that also provide the possibility of continuous monitoring. It has been reported that a training program consisting of six hours may enable physicians who are unexperienced in the field of echocardiography to apply this new method. Up to now, there is no evidence whether this methods is associated with improved postoperative outcome.

Therefore we hypothesize that continuous hemodynamically focussed transesophageal echocardiography positively influences patient outcome (primary hypothesis). Furthermore, its application may decrease hospital expenses (secondary hypothesis).

ELIGIBILITY:
Inclusion Criteria:

* elective, cardiac surgery
* hemodynamic instability or placement of hTEE/PICCO (Pulse Contour Continuous Cardiac Output) /PAC (Pulmonary Arterial Catheter) within 12 hours of ICU admission

Exclusion Criteria:

* pregnant/breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery followed by postoperative observation on an ICU of the anaesthesiology department of the Charité hospital
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Cumulative dosage of catecholamine application | three days beginning upon placement of device

SECONDARY OUTCOMES:
degree and duration of other vasoactive substances | degree and duration of other vasoactive substances three days beginning upon placement of device (or icu admission in control patients, respectively)
  i.e. epinephrine, levosimendan, dopamine, nitroglycerine, nitroprusside
fluid balance | day 1, 2 and 3, beginning upon placement of device (or icu admission in control patients, respectively)
degree and duration of lactate acidosis | degree and duration of other vasoactive substances three days beginning upon placement of device (or icu admission in control patients, respectively)
  maximum lactate level, date/time of maximum lactate level, first date/time when lactate <20
duration of postoperative ventilation | first postoperative day until extubation (2 days on average)
incidence of renal failure | three days beginning upon placement of device (or icu admission in control patients, respectively)
  analysis of creatinine plasma level
incidence of hemodialysis | three days beginning upon placement of device (or icu admission in control patients, respectively)
length of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
in-hospital mortality | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
cost of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Cheitlin MD, Armstrong WF, Aurigemma GP, Beller GA, Bierman FZ, Davis JL, Douglas PS, Faxon DP, Gillam LD, Kimball TR, Kussmaul WG, Pearlman AS, Philbrick JT, Rakowski H, Thys DM, Antman EM, Smith SC Jr, Alpert JS, Gregoratos G, Anderson JL, Hiratzka LF, Faxon DP, Hunt SA, Fuster V, Jacobs AK, Gibbons RJ, Russell RO; ACC; AHA; ASE. ACC/AHA/ASE 2003 Guideline Update for the Clinical Application of Echocardiography: summary article. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/ASE Committee to Update the 1997 Guidelines for the Clinical Application of Echocardiography). J Am Soc Echocardiogr. 2003 Oct;16(10):1091-110. doi: 10.1016/S0894-7317(03)00685-0. No abstract available. PMID 14566308
- [Background] Pearse R, Dawson D, Fawcett J, Rhodes A, Grounds RM, Bennett ED. Early goal-directed therapy after major surgery reduces complications and duration of hospital stay. A randomised, controlled trial [ISRCTN38797445]. Crit Care. 2005;9(6):R687-93. doi: 10.1186/cc3887. Epub 2005 Nov 8. PMID 16356219
- [Background] Giglio MT, Marucci M, Testini M, Brienza N. Goal-directed haemodynamic therapy and gastrointestinal complications in major surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Nov;103(5):637-46. doi: 10.1093/bja/aep279. PMID 19837807
- [Background] Hamilton MA, Cecconi M, Rhodes A. A systematic review and meta-analysis on the use of preemptive hemodynamic intervention to improve postoperative outcomes in moderate and high-risk surgical patients. Anesth Analg. 2011 Jun;112(6):1392-402. doi: 10.1213/ANE.0b013e3181eeaae5. Epub 2010 Oct 21. PMID 20966436
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Background] Futier E, Constantin JM, Petit A, Chanques G, Kwiatkowski F, Flamein R, Slim K, Sapin V, Jaber S, Bazin JE. Conservative vs restrictive individualized goal-directed fluid replacement strategy in major abdominal surgery: A prospective randomized trial. Arch Surg. 2010 Dec;145(12):1193-200. doi: 10.1001/archsurg.2010.275. PMID 21173294
- [Background] Dalfino L, Giglio MT, Puntillo F, Marucci M, Brienza N. Haemodynamic goal-directed therapy and postoperative infections: earlier is better. A systematic review and meta-analysis. Crit Care. 2011 Jun 24;15(3):R154. doi: 10.1186/cc10284. PMID 21702945
- [Background] Grocott MPW, Mythen MG, Gan TJ. Perioperative fluid management and clinical outcomes in adults. Anesth Analg. 2005 Apr;100(4):1093-1106. doi: 10.1213/01.ANE.0000148691.33690.AC. PMID 15781528
- [Background] Vincent JL, Rhodes A, Perel A, Martin GS, Della Rocca G, Vallet B, Pinsky MR, Hofer CK, Teboul JL, de Boode WP, Scolletta S, Vieillard-Baron A, De Backer D, Walley KR, Maggiorini M, Singer M. Clinical review: Update on hemodynamic monitoring--a consensus of 16. Crit Care. 2011 Aug 18;15(4):229. doi: 10.1186/cc10291. PMID 21884645
- [Background] Benjamin E, Griffin K, Leibowitz AB, Manasia A, Oropello JM, Geffroy V, DelGiudice R, Hufanda J, Rosen S, Goldman M. Goal-directed transesophageal echocardiography performed by intensivists to assess left ventricular function: comparison with pulmonary artery catheterization. J Cardiothorac Vasc Anesth. 1998 Feb;12(1):10-5. doi: 10.1016/s1053-0770(98)90048-9. PMID 9509350